CLINICAL TRIAL: NCT02031822
Title: Evaluation of Two Ultrasound-guided Techniques for Greater Occipital Nerve Injections of Local Anesthetic and Steroid for Treatment of Primary Headaches
Brief Title: Two US-guided Techniques for Greater Occipital Nerve Blocks
Acronym: GON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-6804
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2017-10

CONDITIONS: Primary Headache
Keywords: Primary Headache; Greater Occipital Nerve; Ultrasound; Chronic Pain; Cervicogenic; Occipital Neuralgia; Migraine; Tension type headache; Cluster headache
MeSH Terms: conditions — Chronic Pain; Migraine Disorders; Tension-Type Headache; Cluster Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- US-guided Distal GON Block (Group D) (Active Comparator): Needle placement for 2ml 0.5% bupivacaine with epinephrine 1:200,000 and Depo-Medrol 40mg will be performed under US guidance at the level of the superior nuchal line lateral to the external occipital protuberance, close to the occipital artery.
  Interventions: Procedure: US-guided Greater Occipital Nerve Injection
- US-guided Proximal GON Block (Group P) (Active Comparator): Needle placement for 2ml 0.5% bupivacaine with epinephrine 1:200,000 and Depo-Medrol 40mg will be performed under US guidance at the level of the bifid C2 spinous process laterally, between the inferior obliquus capitis and semispinalis capitis muscles.
  Interventions: Procedure: US-guided Greater Occipital Nerve Injection

INTERVENTIONS:
Procedure: US-guided Greater Occipital Nerve Injection — Medication injected around the greater occipital nerve: 2ml 0.5% bupivacaine with epinephrine 1:200,000 and Depo-Medrol 40mg.

SUMMARY:
Headache is one of the most common reasons for patients to access healthcare. Greater occipital nerve (GON) block with local anesthetic and steroid has been described for the management of primary headache refractory to conventional treatment. Two ultrasound (US)-guided techniques for greater occipital nerve (GON) block have been described for the management of refractory headache syndromes: a proximal technique performed at the level of the second cervical vertebra and a distal technique performed at the level of the superior nuchal line. Our airm is to compare the accuracy, efficacy and safety of these two techniques in patients with refractory headaches.

DETAILED DESCRIPTION:
We conducted a double-blinded, randomized control trial to compare accuracy, efficacy and safety of these two techniques in patients with refractory headache syndromes. Following REB approval, 40 patients with moderate or severe refractory headaches (intensity score>4/10) will be randomized to the "proximal" or "distal" groups with a 1:1 allocation. Each patient receives an injection of 2ml of 0.5% bupivacaine with 40mg of methylprednisolone. The null hypothesis is that there is no difference in intensity scores for headache at one month after the interventions. Outcomes related to efficacy (numbness immediately after the injection, reduction in episodes of severe headache, sleep quality), performance (time taken for and discomfort during procedure), and safety (incidence of hematoma, intravascular injection) are measured after one month.

ELIGIBILITY:
Inclusion Criteria:

1. Features suggestive of occipital neuralgia: pain that begins in the upper neck and back of the head with radiation forward toward the eye and has an aching or burning character.
2. Diagnosis of refractory primary headache, any type
3. Baseline NRS headache score of > 4 refractory to conventional oral analgesic therapy (anti-inflammatory drugs, migraine prophylaxis and treatment drugs, opioids).

Exclusion Criteria:

1. Ongoing litigation issues related to the patient's pain
2. Pregnancy
3. Allergy to steroids or local anesthetics
4. Multiple serious comorbidities
5. Age < 18 or age ≥ 80 years
6. GON injection within last 3 months at time of entry into the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2017-09 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Numerical rating score (NRS) for headaches | One month

SECONDARY OUTCOMES:
Efficacy-Related Outcomes | 24 hours and 3 months
  This would include NRS for headache at 24 hrs and 3 months after the intervention, patient satisfaction with the block, Hospital Anxiety and Depression Scale at 1 month compared to baseline, SF-36 Short Form Health Survey to measure improvement in functional status compared to baseline, quality of sleep and average hours of restful sleep at night.
Performance-Related Outcomes | During procedure
  We will measure performance time from contact of US probe with skin to the end of the procedure, procedural discomfort as rated by NRS, number of needle re-adjustments and evidence of sensory block as confirmed by the loss of pin-prick sensation in the dermatomal distribution of GON, and visualization of GON.
Safety-Related Outcomes | Immediate post-procedure and at 1 month
  Any immediate post intervention complications will be recorded (e.g. hematoma, vascular puncture, dizziness). Occurrence of any long-term adverse effects (e.g. infection, numbness, alopecia) will be recorded at 1 month following the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Bhatia, MD FRCPC, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Western Hospital, University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flamer D, Alakkad H, Soneji N, Tumber P, Peng P, Kara J, Hoydonckx Y, Bhatia A. Comparison of two ultrasound-guided techniques for greater occipital nerve injections in chronic migraine: a double-blind, randomized, controlled trial. Reg Anesth Pain Med. 2019 May;44(5):595-603. doi: 10.1136/rapm-2018-100306. Epub 2019 Mar 18. PMID 30886069